CLINICAL TRIAL: NCT04049669
Title: Phase 2 Trial of Indoximod With Chemotherapy and Radiation for Children With Progressive Brain Tumors or Newly Diagnosed DIPG
Brief Title: Pediatric Trial of Indoximod With Chemotherapy and Radiation for Relapsed Brain Tumors or Newly Diagnosed DIPG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Theodore S. Johnson (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Augusta University (Other); Emory University (Other)
Responsible Party: Sponsor-Investigator, Theodore S. Johnson, Associate Professor, Augusta University
Organization: Augusta University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GCC1949; R01CA229646 (NIH)
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; Medulloblastoma; Ependymoma; Diffuse Intrinsic Pontine Glioma
Keywords: IDO; indoleamine 2,3-dioxygenase; indoximod; pediatric; childhood; brain tumor; glioblastoma; medulloblastoma; ependymoma; diffuse intrinsic pontine glioma; DIPG; radiation; temozolomide; cyclophosphamide; etoposide; lomustine; immunotherapy; immune; central nervous system; CNS
MeSH Terms: conditions — Glioblastoma; Medulloblastoma; Ependymoma; Diffuse Intrinsic Pontine Glioma; Brain Neoplasms | interventions — 1-methyltryptophan; Temozolomide; Cyclophosphamide; Etoposide; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Core Regimen, sub-cohort A (Experimental): For patients not eligible for re-irradiation; Start with Core Regimen chemo-immunotherapy (indoximod with oral temozolomide).
  Interventions: Drug: Indoximod; Drug: Temozolomide
- Core Regimen, sub-cohort B (Experimental): For patients who are eligible for partial re-irradiation; Start with indoximod plus up-front re-irradiation, using a palliative low-dose or partial-field radiation plan (low-dose radiation or not all disease sites included); Followed by Core Regimen chemo-immunotherapy (indoximod with oral temozolomide).
  Interventions: Drug: Indoximod; Radiation: Partial Radiation; Drug: Temozolomide
- Core Regimen, sub-cohort C (Experimental): For patients who are eligible for full-dose radiation; (All newly diagnosed DIPG patients and some relapsed ependymoma patients); Start with indoximod plus up-front radiation, using a palliative full-dose radiation plan to all known sites of disease (>50 Gy to brain, >45 Gy to spine); Followed by Core Regimen chemo-immunotherapy (indoximod with oral temozolomide).
  Interventions: Drug: Indoximod; Radiation: Full-dose Radiation; Drug: Temozolomide
- Salvage Regimen 1 (Experimental): For patients who wish to continue access to indoximod after progression on the Core Regimen; Cross-over to indoximod with oral metronomic cyclophosphamide and etoposide).
  Interventions: Drug: Indoximod; Drug: Cyclophosphamide; Drug: Etoposide
- Salvage Regimen 2 (Experimental): For patients who wish to continue access to indoximod after progression on the Core Regimen; Cross-over to indoximod with oral lomustine and temozolomide).
  Interventions: Drug: Indoximod; Drug: Temozolomide; Drug: Lomustine

INTERVENTIONS:
Drug: Indoximod — Indoximod will be taken by mouth twice daily during radiation and throughout each chemo-immunotherapy treatment cycle.
Radiation: Partial Radiation — Palliative low-dose or partial-field radiation plan (low-dose radiation or not all disease sites included).
  Arms: Core Regimen, sub-cohort B
Radiation: Full-dose Radiation — Palliative full-dose radiation plan to all known sites of disease (>50 Gy to brain, >45 Gy to spine).
  Arms: Core Regimen, sub-cohort C
Drug: Temozolomide — Temozolomide will be taken by mouth once daily, on days 1-5 of each chemo-immunotherapy treatment cycle.
  Arms: Core Regimen, sub-cohort A; Core Regimen, sub-cohort B; Core Regimen, sub-cohort C; Salvage Regimen 2
Drug: Cyclophosphamide — Cyclophosphamide will be taken by mouth once daily, on days 1-21 of each chemo-immunotherapy treatment cycle.
  Arms: Salvage Regimen 1
Drug: Etoposide — Etoposide will be taken by mouth once daily, on days 1-21 of each chemo-immunotherapy treatment cycle.
  Arms: Salvage Regimen 1
Drug: Lomustine — Lomustine will be taken by mouth once daily, on day 1 of each chemo-immunotherapy treatment cycle.
  Arms: Salvage Regimen 2

SUMMARY:
Indoximod was developed to inhibit the IDO (indoleamine 2,3-dioxygenase) enzymatic pathway, which is important in the natural regulation of immune responses. This potent immune suppressive mechanism has been implicated in regulating immune responses in settings as diverse as infection, tissue/organ transplant, autoimmunity, and cancer. By inhibiting the IDO pathway, we hypothesize that indoximod will improve antitumor immune responses and thereby slow the growth of tumors.

The central clinical hypothesis for the GCC1949 study is that inhibiting the pivotal IDO pathway by adding indoximod immunotherapy during chemotherapy and/or radiation is a potent approach for breaking immune tolerance to pediatric tumors that will improve outcomes, relative to standard therapy alone.

This is an NCI-funded (R01 CA229646, MPI: Johnson and Munn) open-label phase 2 trial using indoximod-based combination chemo-radio-immunotherapy for treatment of patients age 3 to 21 years who have progressive brain cancer (glioblastoma, medulloblastoma, or ependymoma), or newly-diagnosed diffuse intrinsic pontine glioma (DIPG). Statistical analysis will stratify patients based on whether their treatment plan includes up-front radiation (or proton) therapy in combination with indoximod. Central review of tissue diagnosis from prior surgery is required, except non-biopsied DIPG. This study will use the "immune-adapted Response Assessment for Neuro-Oncology" (iRANO) criteria for measurement of outcomes. Planned enrollment is up to 140 patients.

DETAILED DESCRIPTION:
Disease-specific Cohorts :

Cohort 1A, 1B (closed to enrollment): relapsed or refractory glioblastoma

Cohort 2A, 2B: relapsed or refractory medulloblastoma

Cohort 3A, 3B, 3C: relapsed or refractory ependymoma

Cohort 4C (closed to enrollment): newly-diagnosed DIPG (must have no prior radiation or other therapy)

.

Radiation (or proton) plan sub-cohorts:

Sub-cohort A: for patients not eligible for re-irradiation

Sub-cohort B: for patients who are eligible for partial re-irradiation

Sub-cohort C: for patients who are eligible for full-dose radiation (All newly diagnosed DIPG patients and some relapsed ependymoma patients)

ELIGIBILITY:
Inclusion Criteria:

Diagnosis:

* Progressive disease with histologically proven initial diagnosis of glioblastoma, medulloblastoma, or ependymoma; With confirmation of progression by either MRI or CSF analysis; Measureable disease is not required for study entry; Patients with progressive disease must have been previously treated with therapeutic radiation as part of treatment for the initial brain cancer diagnosis or for a prior relapse.
* Newly diagnosed DIPG (diffuse intrinsic pontine glioma) with no prior therapy (including no prior radiation); Biopsy is not required for DIPG.
* Central review of tissue diagnosis is required, except non-biopsied DIPG; Archival tumor tissue must be located and available prior to study entry.
* Patients with metastatic disease are eligible.

Lansky or Karnofsky performance status score must be ≥ 50%.

Adequate renal function: creatinine ≤ 1.5-times upper limit of age-adjusted normal.

Adequate liver function:

* ALT ≤ 5-times upper limit of normal.
* Total bilirubin ≤ 1.5-times upper limit of normal.

Adequate Bone marrow function:

* Absolute neutrophil count (ANC) ≥ 750/mcL.
* Platelets ≥ 75,000/mcL (transfusion independent).
* Hemoglobin ≥ 8 g/dL (transfusion independent).

Central nervous system: seizure disorders must be well controlled on antiepileptic medication.

Prior therapy

* DIPG patients must not have been treated with any prior radiation or medical therapy.
* Patients previously treated with indoximod are excluded.
* Patients previously treated with any other immunotherapy agent, including other IDO-targeted drugs, are eligible for enrollment.
* Patients previously treated with chemotherapy drugs included in this protocol are eligible for enrollment.

Patients must be 14 days from the administration of any investigational agent or prior cytotoxic therapy with the following exceptions:

* Temozolomide dosed at or above 150 mg/m2 (allowed, but must be at least 21 days from the last dose of temozolomide).
* Must be 28 days from administration of antibody-based therapies (e.g., bevacizumab), tumor-directed vaccines, or cellular immune therapies (e.g., T cells, NK cells, etc).
* Must be 56 days from administration of tumor-directed therapies using infectious agents (e.g., viruses, bacteria, etc).

Pregnant women are excluded from this study, where pregnancy is confirmed by a positive urine or serum hCG laboratory test.

Patients must be able to swallow pills.

.

Exclusion Criteria:

Patients who cannot swallow indoximod pills are excluded.

Patients previously treated with indoximod are excluded.

Patients with DIPG who have been treated with any prior radiation or medical therapy are excluded.

Midline glioma that does not include significant brain stem involvement is not considered DIPG for enrollment purposes, and is excluded.

Patients with active systemic infection requiring treatment, including any HIV infection or toxoplasmosis, are excluded.

Patients with active autoimmune disease that requires systemic therapy are excluded.

Pregnant women are excluded

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2027-10-02 (Estimated)

PRIMARY OUTCOMES:
8-month iRANO-PFS (Progression-Free Survival, defined by immune-adapted iRANO criteria) | Up to 5 years
  For patients with relapsed glioblastoma, medulloblastoma, or ependymoma.
12-month Overall Survival (OS) | Up to 5 years
  For patients with newly diagnosed DIPG (diffuse intrinsic pontine glioma).

SECONDARY OUTCOMES:
Median Overall Survival (OS) | Up to 5 years
  For each disease cohort
Median iRANO-PFS (Progression-Free Survival, defined by immune-adapted iRANO criteria) | Up to 5 years
  For each disease cohort
Median Time to Regimen Failure (TTRF) | Up to 5 years
  For each disease cohort

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S Johnson, MD, PhD, Principal Investigator — Augusta University
Locations (5):
- United States (5):
  - Augusta University, Georgia Cancer Center, Augusta, Georgia
  - Emory University, Children's Heathcare of Atlanta, Druid Hills, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Johnson TS, MacDonald TJ, Pacholczyk R, Aguilera D, Al-Basheer A, Bajaj M, Bandopadhayay P, Berrong Z, Bouffet E, Castellino RC, Dorris K, Eaton BR, Esiashvili N, Fangusaro JR, Foreman N, Fridlyand D, Giller C, Heger IM, Huang C, Kadom N, Kennedy EP, Manoharan N, Martin W, McDonough C, Parker RS, Ramaswamy V, Ring E, Rojiani A, Sadek RF, Satpathy S, Schniederjan M, Smith A, Smith C, Thomas BE, Vaizer R, Yeo KK, Bhasin MK, Munn DH. Indoximod-based chemo-immunotherapy for pediatric brain tumors: A first-in-children phase I trial. Neuro Oncol. 2024 Feb 2;26(2):348-361. doi: 10.1093/neuonc/noad174. PMID 37715730
- [Background] Sharma MD, Pacholczyk R, Shi H, Berrong ZJ, Zakharia Y, Greco A, Chang CS, Eathiraj S, Kennedy E, Cash T, Bollag RJ, Kolhe R, Sadek R, McGaha TL, Rodriguez P, Mandula J, Blazar BR, Johnson TS, Munn DH. Inhibition of the BTK-IDO-mTOR axis promotes differentiation of monocyte-lineage dendritic cells and enhances anti-tumor T cell immunity. Immunity. 2021 Oct 12;54(10):2354-2371.e8. doi: 10.1016/j.immuni.2021.09.005. Epub 2021 Oct 5. PMID 34614413